CLINICAL TRIAL: NCT01833065
Title: A Double-blind, Randomised, Placebo-controlled, Phase 3 Trial in Patients With Chronic Idiopathic Constipation to Demonstrate the Efficacy and Safety of Elobixibat 5 mg and 10 mg for 12 Weeks Followed by a 4-week Withdrawal Period
Brief Title: Efficacy and Safety Trial of Elobixibat in Patients With Chronic Idiopathic Constipation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to a distribution issue with the trial medication
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000080; 2012-005588-28 (EudraCT Number)
Record Dates: First submitted 2013-04-12; First posted 2013-04-16 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — elobixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EBX 10 (Experimental): Elobixibat 10 mg/day
  Interventions: Drug: Elobixibat 10 mg/day
- EBX 5 (Experimental): Elobixibat 5 mg/day
  Interventions: Drug: Elobixibat 5 mg/day
- PLCBO (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elobixibat 10 mg/day — Elobixibat 10 mg/day
  Other Names: A3309
  Arms: EBX 10
Drug: Elobixibat 5 mg/day — Elobixibat 5 mg/day
  Other Names: A3309
  Arms: EBX 5
Drug: Placebo — Placebo
  Arms: PLCBO

SUMMARY:
12 Week Efficacy and Safety Trial Followed by a 4 Week Withdrawal Period for Patients with Chronic Idiopathic Constipation.

DETAILED DESCRIPTION:
The present trial was designed to determine the efficacy and safety of elobixibat treatment (at both doses of 5 mg and 10 mg/day) compared to placebo treatment for 12-week Treatment Period followed by a 4-week Withdrawal Period in patients with chronic idiopathic constipation. During Withdrawal Period a sub-group of patients in elobixibat 5 mg and 10 mg treatment arms respectively received placebo treatment, while rest of the patients continued with 5 mg and 10 mg treatment in respective groups. In placebo groups, patients received elobixibat 10 mg treatment during Withdrawal Period. Patients were followed-up for 2 weeks after end of the Withdrawal Period.

The assessment of primary and key secondary end points was done for patients who completed the first 12 weeks of treatment period. Incidence of Adverse Events (AEs) were reported till 2 weeks after end of the Withdrawal Period.

The trial was early terminated due to a distribution issue with the trial medication.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.5 but <35.0 kg/m^2
* Male or female ≥18 years of age
* Reports <3 spontaneous Bowel Movements (BM) per week and reports one or more of the following symptoms for the last 3 months with symptom onset at least 6 months before the Screening Visit or before starting chronic therapy with any laxative:

  1. Straining during at least 25% of defecations
  2. Lumpy or hard stools during at least 25% of defecations
  3. Sensation of incomplete evacuation during at least 25% of defecations
* Is ambulatory and community dwelling
* An initial colonoscopy is required if recommended by national guidelines

Exclusion Criteria:

* Reports loose (mushy) or watery stools in the absence of any laxative intake in the form of a tablet, a suppository or an enema, or prohibited medicine for >25% of BMs
* The patient reports a BSFS of 6 or 7 during the Pretreatment Period
* Has irritable bowel syndrome (IBS) with pain/discomfort as predominant symptoms
* Has a structural abnormality of the Gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Has a history of diverticulitis, chronic pancreatitis, active peptic ulcer disease (PUD) not adequately treated, ischaemic colitis, inflammatory bowel disease, laxative abuse, faecal impaction that required hospitalization or emergency treatment, pseudo-obstruction, megacolon, megarectum, bowel obstruction, descending perineum syndrome, ovarian cysts, endometriosis, solitary rectal ulcer syndrome, systemic sclerosis, pre-malignant colonic disease (e.g., familial adenomatous polyposis or hereditary non-polyposis colorectal cancer) or other forms of familial colorectal cancer
* Has unexplained and clinically significant GI alarm signals (e.g., lower GI bleeding or heme-positive stool in the absence of known internal or external haemorrhoids, iron-deficiency anaemia, unexplained weight loss) or systemic signs of infection or colitis
* Has a potential central nervous system (CNS) cause of constipation (e.g., Parkinson's disease, spinal cord injury, multiple sclerosis)
* Has intestinal/rectal prolapse or other known pelvic floor dysfunction
* Commonly uses digital maneuvers (perianal pressure or digital disimpaction) or vaginal splinting to facilitate the passage of a bowel movement
* Has a history of diabetic neuropathy
* Has a history of bariatric surgery for treatment of obesity; surgery to remove a segment of the GI tract; or surgery of the abdomen, pelvic or retroperitoneal area during the 6 months prior to Screening; or appendectomy or cholecystectomy 3 months prior to screening; or other major surgery 1 month prior to Screening
* Has a history of cancer with last date of proven disease activity/presence of malignancy within 5 years, except for adequately treated basal cell carcinoma of the skin, cervical dysplasia, or carcinoma in situ of the skin or the cervix
* Known human immunodeficiency virus (HIV) or Hepatitis B/C (HBV/HCV) infection
* Has a history of hospitalization for any psychiatric disorder, or any suicide attempt in the 2 years prior to Screening
* Is actively abusing alcohol or drugs or has a history of alcohol or drug abuse during the 6 months prior to Screening
* Is being treated for hypothyroidism, but the dose of medication has not been stable for at least 3 months at the time of Screening
* Is a pregnant, breast-feeding, or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (97):
- United States (45):
  - Birmingham Gastroenterology Associates, PC, Birmingham, Alabama
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - David Geffen School of Medicine at University of California, Los Angeles, Los Angeles, California
  - West Gastroenterology Associates, Los Angeles, California
  - Sacramento Research Medical Group, Sacramento, California
  - Precision Research Institute, LLC, San Diego, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Zasa Clinical Research, Boynton Beach, Florida
  - Meridien Research, Bradenton, Florida
  - Sanitas Research, Coral Gables, Florida
  - Lake Internal Medicine Associates, Eustis, Florida
  - Health Care Family Rehab Corp., Hialeah, Florida
  - Southeast Clinical Research, LLC, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - Premier Healthcare Research, LLC, Evanston, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Professional Research Network of Kansas, LLC, Witchita, Kansas
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Carolina Digestive Health Associates, PA, Charlotte, North Carolina
  - Carolina Digestive Health Associates, PA, Concord, North Carolina
  - PharmQuest, LLC, Greensboro, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Hometown Urgent Care and Occupational Health, Columbus, Ohio
  - Hometown Urgent Care and Occupational Health, Dayton, Ohio
  - Family Practice Center of Wadsworth, Wadsworth, Ohio
  - Clinical Research Associates, LLC, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Family Medical Associates, Levittown, Pennsylvania
  - Anderson Gastroenterology Associates, Anderson, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Associates in Gastroenterology, LLC, Hermitage, Tennessee
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - New Phase Research and Development, LLC, Knoxville, Tennessee
  - Research Across America, Katy, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
- Brazil (3):
  - Fundacao IMEPEM - Universidade Federal de Juiz de Fora, Juiz de Fora, Minas Gerais
  - Gastrocentro Carioca Centro Gast e Endosc Dig, Ltda, Rio de Janeiro, Rio de Janeiro
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
- Canada (5):
  - Medical Arts Health Research Group, Penticton, British Columbia
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Dr Anil K Gupta Medicine Professional Corp., Toronto, Ontario
  - Toronto Digestive Diseases Associates, Inc., Toronto, Ontario
  - Pro-Recherche Polyclinique des Ponts, Saint Romuald, Quebec
- Czechia (2):
  - Fakultní Nemocnice Ostrava, Ostrava, Severomoravsky Kraj
  - Gastroenterologicka a interni ambulance, České Budějovice
- Germany (3):
  - Synexus Clinical Research GmbH, Dresden, Saxony
  - Synexus Clinical Research GmbH, Görlitz, Saxony
  - Synexus Clinical Research GmbH, Magdeburg, Saxony-Anhalt
- Hungary (10):
  - Pándy Kálmán Megyei Kórház, Gyula, Bekes County
  - Jahn Ferenc Dél-Pesti Kórház és Rendelointézet, Budapest
  - Pannónia Magánorvosi Centrum Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Vasútegészségügyi Nonprofit Kiemelten Közhasznú Kft, Debrecen
  - Borsod Abaúj Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Miskolci Semmelweis Kórház és Egyetemi Oktatókórház, Miskolc
  - Clinfan Szolgáltató Kft, Szekszárd
  - CRU Hungary Kft., Szikszó
  - Jávorszky Ödön Kórház, Vác
- Mexico (4):
  - Hospital Centro Internacional de Medicina Chihuahua, Chihuahua City, Chihuahua
  - Centro de Investigación Médico Biológica y Terapia Avanzada SC, Guadalajara, Jalisco
  - Accelerium Clinical Research, Monterrey, Nuevo León
  - Medical Care and Research, Mérida, Yucatán
- Poland (7):
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska Adam Kopon, Torun, Kuyavian-Pomeranian Voivodeship
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Medica Pro Familia Sp. z o.o. S.K.A., Warsaw, Masovian Voivodeship
  - Przychodnia Polskiej Fundacji Gastroenterologii Filia Nr 1 NZOZ, Warsaw, Masovian Voivodeship
  - Medicor Centrum Medyczne Tadeusz Mazurek, Rzeszów, Podkarpackie Voivodeship
  - SPZOZ Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lódz, Łódź Voivodeship
- Slovakia (5):
  - Gastro I.s.r.o., Prešov, Presov
  - Lama Medical Care s.r.o., Gastroentero-hepatologicke centrum Thalion, Bratislava
  - PIGEAS s.r.o., Martin
  - KM Management sro, Nitra
  - GEA s.r.o Gastroenterologicka ambulancia, Trnava
- South Africa (6):
  - JOSHA Research, Bloemfontein, Free State
  - Synexus Clinical Research SA, Pretoria, Gauteng
  - Dr. Zubar Fazel Vawda, Durban, KwaZulu-Natal
  - Mzansi Ethical Research Centre, Middelburg, Mpumalanga
  - Louis Leipoldt Medi-Clinic Medical Centre, Bellville, Western Cape
  - Be Part Yoluntu Centre, Paarl, Western Cape
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital Huddinge, Stockholm
  - Uppsala Akademiska Sjukhus, Uppsala
- United Kingdom (4):
  - Synexus Lancashire Clinical Research Centre, Chorley, England
  - Synexus Merseyside Clinical Research Centre, Liverpool, England
  - Synexus Thames Valley Clinical Research Centre, Reading, England
  - Synexus Scotland Clinical Research Centre, Glasgow, Scotland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Trial included 4-week Screening and 2-week Pretreatment Period before patient randomization to treatment sequences i.e. EBX 10/EBX 10, EBX 10/PLCBO, EBX 5/EBX 5, EBX 5/PLCBO and PLCBO/EBX 10. The total study duration was of 16 weeks: the efficacy assessments focused on the first 12 weeks, while safety assessments focused on whole 16 weeks
Groups:
- EBX 10/EBX 10: Patients in this arm received Elobixibat 10 mg/day during the 12-week Treatment Period (i.e. 12 week efficacy assessment) and also received Elobixibat 10 mg/day during the 4-week Withdrawal Period (i.e. 16 week safety assessment).
- EBX 10/PLCBO: Patients in this arm received Elobixibat 10 mg/day during the 12-week Treatment Period (i.e. 12 week efficacy assessment) and received placebo during the 4-week Withdrawal Period (i.e. 16 week safety assessment).
- EBX 5/EBX 5: Patients in this arm received Elobixibat 5 mg/day during the 12-week Treatment Period (i.e. 12 week efficacy assessment) and also received Elobixibat 5 mg/day during the 4-week Withdrawal Period (i.e. 16 week safety assessment).
- EBX 5/PLCBO: Patients in this arm received Elobixibat 5 mg/day during the 12-week Treatment Period (i.e. 12 week efficacy assessment) and received placebo during the 4-week Withdrawal Period (i.e. 16 week safety assessment).
- PLCBO/EBX 10: Patients in this arm received placebo during the 12-week Treatment Period (i.e. 12 week efficacy assessment) and received Elobixibat 10 mg/day during the 4-week Withdrawal Period (i.e. 16 week safety assessment).
Period: Overall Study
Arm/Group | EBX 10/EBX 10 | EBX 10/PLCBO | EBX 5/EBX 5 | EBX 5/PLCBO | PLCBO/EBX 10
Started | 65 (Randomized patients - As treated) | 53 (Randomized patients - As treated) | 35 (Randomized patients - As treated) | 50 (Randomized patients - As treated) | 110 (Randomized patients - As treated)
Intention-to-treat Analysis Set | 50 (Randomized patients) | 53 (Randomized patients) | 50 (Randomized patients) | 50 (Randomized patients) | 111 (Randomized patients)
Completed | 41 | 40 | 23 | 41 | 74
Not Completed | 24 | 13 | 12 | 9 | 36
Not completed — Adverse Event | 6 | 1 | 0 | 2 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 6 | 2 | 4 | 3 | 11
Not completed — Subject's substantial non-compliance | 0 | 1 | 0 | 0 | 0
Not completed — Trial terminated by sponsor | 8 | 8 | 7 | 3 | 13
Not completed — Others | 2 | 1 | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) analysis set.
Groups:
- EBX 10: Elobixibat 10 mg/day was administered orally in a tablet form.
- EBX 5: Elobixibat 5 mg/day was administered orally in a tablet form.
- PLCBO: Placebo was administered orally in a tablet form.
- Total: Total of all reporting groups
Arm/Group | EBX 10 | EBX 5 | PLCBO | Total
Number analyzed (Participants) | 103 | 100 | 111 | 314
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.6 (14.3) | 49.5 (13.5) | 48.0 (16.1) | 49.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 85 | 97 | 266
  Male | 19 | 15 | 14 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 11 | 29
  Not Hispanic or Latino | 94 | 91 | 100 | 285
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 13 | 16 | 45
  White | 85 | 86 | 93 | 264
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 2 | 1 | 4
  Czech Republic | 2 | 2 | 0 | 4
  Sweden | 1 | 2 | 3 | 6
  Hungary | 15 | 13 | 14 | 42
  United States | 49 | 54 | 55 | 158
  Poland | 3 | 4 | 3 | 10
  South Africa | 12 | 7 | 13 | 32
  United Kingdom | 11 | 9 | 12 | 32
  Slovakia | 5 | 3 | 5 | 13
  Germany | 4 | 4 | 5 | 13
Weekly number of CSBM [Mean (Standard Deviation); unit: CSBM per week] — CSBM was defined as a spontaneous (occurring without laxative within the preceding 24 hours, including no rescue medication within the preceding 24 hours) bowel movement (as interpreted by the patient, with a beginning and an end, including single or multiple stools), accompanied by a patient reported sense of complete evacuation ('complete').
  Baseline value for the number of CSBM per week was defined as the average of the numbers of CSBM per week for over the 2-week Pretreatment Period.
  CSBM per week | 0.33 (0.62) | 0.32 (0.62) | 0.43 (0.68) | 0.36 (0.64)
Weekly number of SBM [Mean (Standard Deviation); unit: SBM per week] — SBM was defined as a bowel movement that occurred in the absence of a laxative use or manual disimpaction.
  Baseline value for the number of SBM was defined as the average of the numbers of SBM per week for over the 2-week Pretreatment Period.
  SBM per week | 2.31 (1.27) | 2.19 (1.13) | 2.45 (1.35) | 2.32 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Overall Complete Spontaneous Bowel Movement (CSBM) Response
Description: This outcome measured the percentage of patients who were CSBM responders. A CSBM responder was defined as a patient with ≥3 CSBMs per week and an increase of ≥1 CSBM per week from Baseline, for at least 9 of the 12 weeks in the 12-week Treatment Period, including at least 3 weeks during Weeks 9-12.
Time Frame: During the first 12 weeks
Population: The ITT analysis set consisting of all randomized (as planned) patients.
Measure: Number; unit: Percentage of patients
Groups:
- EBX 10: Elobixibat 10 mg/day was administered orally in a tablet form starting from Baseline visit till end of 12-week Treatment Period.
- EBX 5: Elobixibat 5 mg/day was administered orally in a tablet form starting from Baseline visit till end of 12-week Treatment Period.
- PLCBO: Placebo was administered orally in a tablet form starting from Baseline visit till end of 12-week Treatment Period.
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 103 | 100 | 111
Percentage of patients | 12.6 | 15.0 | 8.1

2. Secondary Outcome: Occurrence of CSBM Response
Description: This outcome measured the percentage of patients who had a CSBM within 24 hours after the first dose of treatment. A CSBM was defined as a spontaneous (occurring without laxative within the preceding 24 hours, including no rescue medication within the preceding 24 hours) bowel movement (as interpreted by the patient, with a beginning and an end, including single or multiple stools), accompanied by a patient reported sense of complete evacuation ('complete').
Time Frame: Within first 24 hours of treatment initiation
Population: The ITT analysis set consisting of all randomized (as planned) patients.
Measure: Number; unit: Percentage of patients
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 103 | 100 | 111
Percentage of patients | 21.4 | 13.0 | 13.5

3. Secondary Outcome: Change From Baseline in Weekly Frequency of Spontaneous Bowel Movement (SBMs)
Description: The change from Baseline for the continuous variable was estimated using a repeated measures analysis of covariance (ANCOVA) model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisting of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: SBM per week
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 103 | 100 | 111
SBM per week | 2.25 [1.78 to 2.71] | 2.40 [1.92 to 2.88] | 1.20 [0.74 to 1.66]

4. Secondary Outcome: Change From Baseline in Weekly Stool Consistency of SBMs
Description: The stool consistency is measured using the seven-point ordinal Bristol Stool Form Scale (BSFS) score. The BSFS classifies human stool into seven types and points them accordingly.
  Type 1: Separate hard lumps, like nuts (hard to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft Type 5: Soft blobs with clear cut edges (passed easily) Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces, entirely liquid Types 1 and 2 indicate constipation, with 3 and 4 represents the ideal stool form (especially the latter), and 5, 6 and 7 tends towards diarrhoea .
  For a given assessment week, the weekly stool consistency was defined as the sum of non-missing stool consistency score for SBMs during that week divided by the number of non-missing stool consistency score for SBMs during that week. The parameter was analysed using repeated measures ANCOVA model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisting of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on BSFS
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 103 | 100 | 111
Units on BSFS | 1.56 [1.35 to 1.77] | 1.45 [1.24 to 1.66] | 0.80 [0.60 to 1.00]

5. Secondary Outcome: Total Patient Assessment of Constipation - Quality of Life (PAC-QOL) Score Responder
Description: This outcome measured the percentage of patients who were PAC-QOL score responder at 12-week Treatment Period. A PAC-QOL score responder was defined as a patient with ≥50% reduction in total PAC-QOL score from Baseline at Week 12.
  PAC-QOL is a 28-item questionnaire for psychometric assessment of disease-specific quality of life. The questionnaire is based on 5-point Likert scale; ranging from 0 [none of the time or not at all] to 4 [all of the time or extremely]). A lower score indicates a better Quality of Life. The PAC-QOL questionnaire is developed specifically for patients with constipation.
  Total PAC-QOL score was averaged from the individual item score.
Time Frame: At Week 12
Population: The ITT analysis set consisting of all randomized (as planned) patients.
Measure: Number; unit: Percentage of patients
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 103 | 100 | 111
Percentage of patients | 33.0 | 31.0 | 18.9

6. Secondary Outcome: Change From Baseline in Weekly Degree of Straining of SBMs
Description: The degree of straining was measured using the five-point ordinal scale (1=Not at all, 2=A little bit, 3=A moderate amount, 4=A great deal, and 5=An extreme amount).
  For a given assessment week, the weekly degree of straining was defined as the sum of non-missing straining score for SBMs during that week divided by the number of non-missing straining score for SBMs during that week. The parameter was analysed using repeated measures ANCOVA model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisting of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 103 | 100 | 111
Units on a scale | -0.90 [-1.03 to -0.77] | -0.84 [-0.97 to -0.71] | -0.63 [-0.76 to -0.50]

7. Secondary Outcome: Change From Baseline in Weekly Abdominal Bloating Score
Description: The abdominal pain score was measured using the five-point ordinal scale (1=None, 2=Mild, 3=Moderate, 4=Severe, and 5=Very severe).
  For a given assessment week, the weekly abdominal bloating score was defined as the sum of non-missing abdominal bloating score for SBMs during that week divided by the number of non-missing abdominal bloating score for SBMs during that week. The parameter was analysed using repeated measures ANCOVA model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisting of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 103 | 100 | 111
Units on a scale | -0.46 [-0.56 to -0.36] | -0.35 [-0.46 to -0.25] | -0.30 [-0.40 to -0.20]

8. Secondary Outcome: Change From Baseline in Weekly Abdominal Discomfort Score
Description: The abdominal discomfort score was measured using the five-point ordinal scale (1=None, 2=Mild, 3=Moderate, 4=Severe, and 5=Very severe).
  For a given assessment week, the weekly abdominal discomfort score was defined as the sum of non-missing abdominal discomfort score for SBMs during that week divided by the number of non-missing abdominal discomfort score for SBMs during that week. The parameter was analysed using repeated measures ANCOVA model.
Time Frame: From Baseline (2-week Pretreatment Period) to overall first 12-weeks of Treatment Period
Population: The ITT analysis set consisting of all randomized (as planned) patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EBX 10 | EBX 5 | PLCBO
Number analyzed (Participants) | 103 | 100 | 111
Units on a scale | -0.37 [-0.48 to -0.27] | -0.32 [-0.43 to -0.22] | -0.25 [-0.36 to -0.15]

ADVERSE EVENTS:
Time Frame: 6 months
Description: The Investigator monitored the condition of the patient and recorded all AEs throughout the trial from the time of obtaining informed consent until the last visit (i.e. the end of the follow-up period, as applicable) in the AEs Log. Information on AEs was collected at each trial visit.
Groups:
- EBX 10/EBX 10: Patients in this arm received Elobixibat 10 mg/day during the 12-week Treatment Period and also received Elobixibat 10 mg/day during the 4-week Withdrawal Period.
- EBX 10/PLCBO: Patients in this arm received Elobixibat 10 mg/day during the 12-week Treatment Period and received placebo during the 4-week Withdrawal Period.
- EBX 5/EBX 5: Patients in this arm received Elobixibat 5 mg/day during the 12-week Treatment Period and also received Elobixibat 5 mg/day during the 4-week Withdrawal Period.
- EBX 5/PLCBO: Patients in this arm received Elobixibat 5 mg/day during the 12-week Treatment Period and received placebo during the 4-week Withdrawal Period.
- PLCBO/EBX 10: Patients in this arm received placebo during the 12-week Treatment Period and received Elobixibat 10 mg/day during the 4-week Withdrawal Period.
Arm/Group | EBX 10/EBX 10 | EBX 10/PLCBO | EBX 5/EBX 5 | EBX 5/PLCBO | PLCBO/EBX 10
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/53 | 0/35 | 1/50 | 3/110
Other Adverse Events (participants affected / at risk) | 25/65 | 11/53 | 13/35 | 20/50 | 24/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBX 10/EBX 10 (N=65) | EBX 10/PLCBO (N=53) | EBX 5/EBX 5 (N=35) | EBX 5/PLCBO (N=50) | PLCBO/EBX 10 (N=110)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBX 10/EBX 10 (N=65) | EBX 10/PLCBO (N=53) | EBX 5/EBX 5 (N=35) | EBX 5/PLCBO (N=50) | PLCBO/EBX 10 (N=110)
Diarrhoea (Gastrointestinal disorders) | 13 (17) | 2 (12) | 1 (2) | 5 (7) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 3 (3) | 2 (2) | 1 (1) | 6 (9)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 5 (5)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (5) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, outcomes were presented only for descriptive purposes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.